CLINICAL TRIAL: NCT04230122
Title: A Single Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of LY3478006 in Healthy Subjects
Brief Title: A Study of LY3478006 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol stopping criteria (safety) were met.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17458; J2F-MC-OHAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10 milligram (mg) LY3478006 - Intravenous (IV) (Experimental): Participants received single dose of 10 mg LY3478006 administered IV. Due to early termination of the study Cohort 2 to 6 (30 mg, 100 mg, 300 mg, 600 mg, and 1000 mg LY3478006 IV) were not explored for safety reasons following dosing of the first 4 participants in Cohort 1.
  Interventions: Drug: LY3478006 - IV
- Placebo - IV (Placebo Comparator): Participants received single dose of placebo administered IV. Placebo IV Cohorts 2 through 6 were not explored as study was terminated for safety reasons following dosing of the first 4 participants in cohort 1.
  Interventions: Drug: Placebo - IV
- 100 mg LY3478006 - Subcutaneous (SC) (Cohort 7) (Experimental): 100 mg LY3478006 cohort 7 SC dose was not explored as study was terminated for safety reasons following dosing of the first 4 participants in cohort 1.
  Interventions: Drug: LY3478006 - SC
- Placebo - SC (Cohort 7) (Placebo Comparator): Placebo cohort 7 SC dose were not explored as study was terminated for safety reasons following dosing of the first 4 participants in cohort 1.
  Interventions: Drug: Placebo - SC

INTERVENTIONS:
Drug: LY3478006 - IV — Administered IV
  Arms: 10 milligram (mg) LY3478006 - Intravenous (IV)
Drug: LY3478006 - SC — Administered SC
  Arms: 100 mg LY3478006 - Subcutaneous (SC) (Cohort 7)
Drug: Placebo - IV — Administered IV
  Arms: Placebo - IV
Drug: Placebo - SC — Administered SC
  Arms: Placebo - SC (Cohort 7)

SUMMARY:
The purpose of this study is to learn more about how safe and how well tolerated LY3478006 is when given by injection into a vein or just under the skin to healthy participants. Blood tests will be done to check how much LY3478006 is in the bloodstream and how long the body takes to get rid of it. For each participant, the study will last up to about 16 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy male or female Japanese or non-Japanese participants, as determined by medical history and physical examination
* Women not of childbearing potential
* Are aged 18 to 55 years (20 to 55 years for Japanese participants), inclusive, at screening

Exclusion Criteria:

* Have clinically significant abnormal electrocardiogram (ECG) results
* Have persistent abnormal blood pressure or pulse rate, as determined by the investigator
* Have evidence of orthostatic hypotension, defined as a decrease in systolic or diastolic blood pressure greater than or equal to (≥)20 millimeters of mercury (mmHg) or ≥10 mmHg, respectively
* Have significant history or presence of cardiovascular, respiratory, hepatic, ophthalmological, renal, gastrointestinal, endocrine, hematological, neurological, or psychiatric disorders
* Have a history or presence of mononeuropathy, polyneuropathy, or autonomic neuropathy
* Have significant allergies to humanized monoclonal antibodies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 Milligram (mg) LY3478006 - Intravenous (IV): Participants received single dose of 10 mg LY3478006 administered IV.
- Placebo - IV: Participants received single dose of placebo administered IV.
Period: Overall Study
Arm/Group | 10 Milligram (mg) LY3478006 - Intravenous (IV) | Placebo - IV
Started | 3 | 1
Received at Least 1 Dose of Study Drug | 3 | 1
Completed | 2 | 1
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 10 mg LY3478006 - IV: Participants received single dose of 10 mg LY3478006 administered IV.
- Total: Total of all reporting groups
Arm/Group | 10 mg LY3478006 - IV | Placebo - IV | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (10.4) | 33 (NA) — Value was not evaluable because only one participant was analyzed. | 34.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Data presented are the number of participants who experienced SAEs considered by the investigator to be related to study drug administration. A summary of SAEs and all other non-serious Adverse Event(s) (AEs), regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline through study completion (up to 109 days)
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg LY3478006 - IV | Placebo - IV
Number analyzed (Participants) | 3 | 1
Participants | 3 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3478006
Description: Cmax of LY3478006 was evaluated.
Time Frame: Predose; Day 1 with end of infusion, 3, 6, 12 hours
Population: All randomized participants who received at least one dose of study drug and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | 10 mg LY3478006 - IV
Number analyzed (Participants) | 3
microgram per milliliter (μg/mL) | 2.3 (22)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC0-∞) of LY3478006
Description: AUC0-∞ of LY3478006 was evaluated. The unit of measure is hour*microgram per milliliter (hr*mcg/mL).
Time Frame: Predose; Day 1 with end of infusion, 3, 6, 12 hours; Day 2; Day 3; Day 5; Day 8; Day 10; Day 15; Day 22; Day 29; Day 43; Day 57; Day 71 and Day 85
Population: All randomized participants who received at least one dose of study drug and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*mcg/mL
Arm/Group | 10 mg LY3478006 - IV
Number analyzed (Participants) | 3
hr*mcg/mL | 550 (8.03)

ADVERSE EVENTS:
Time Frame: Baseline through study completion (up to 109 days)
Description: All randomized participants who received at least one dose of study drug.
Groups:
- 10 mg LY3478006 IV: Participants received single dose of placebo administered IV.
- Placebo IV: Participants received single dose of 10 mg LY3478006 administered IV.
Arm/Group | 10 mg LY3478006 IV | Placebo IV
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg LY3478006 IV (N=3) | Placebo IV (N=1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0) — One participant SAE was resolved after study completion with resolution occurring on day 138.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg LY3478006 IV (N=3) | Placebo IV (N=1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Cohort 2 through 7 were not explored as study was terminated early for safety reasons after Cohort 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-12-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT04230122/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT04230122/SAP_001.pdf